CLINICAL TRIAL: NCT07310914
Title: Implementation of an Advanced Telerehabilitation Solution for People With Multiple Sclerosis
Acronym: PLATINUMS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Danish Multiple Sclerosis Hospitals (Other)
Collaborators: MS Ireland (Unknown); Tel Aviv University (Other); University of Cagliari (Other); University of Limerick (Other)
Responsible Party: Principal Investigator, Lars Hvid, Senior Researcher, PHD, Danish Multiple Sclerosis Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telerehabilitation in PWMS
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Neurorehabilitation; Telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 10 weeks of home-based exercise performed with the telerehabilitation system. Partipicants will perform two sessions per week (30-45 minutes). The content of the exercise program and the specific exercises will be planned by specialized physiotherapists.
  Interventions: Behavioral: Telerehabilitation
- Paper-based instructions (Active Comparator): 10 weeks of home-based exercise with paper-based instructions. Partipicants will perform two sessions per week (30-45 minutes). The content of the exercise program and the specific exercises will be planned by specialized physiotherapists.Paper-based exercise instructions
  Interventions: Behavioral: Paper-based exercise

INTERVENTIONS:
Behavioral: Telerehabilitation — Advanced telerehabilitation with a program made by specialized physiotherapists and delivered through the WizeCare system.
  Arms: Experimental
Behavioral: Paper-based exercise — Paper-based exercise instructions made by specialized physiotherapists.
  Arms: Paper-based instructions

SUMMARY:
The overall purpose of the present study is to investigate the effect of an advanced telerehablitation system (TRS) in persons with multiple sclerosis on mobility. The advanced telerhabilitation system is based on AI components, and delivers instant feedback to the partcipants. If the project is successful, it can help optimize exercise for those persons with multiple sclerosis who are either not able or willing to travel to a clinical setting for exericse.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of MS according to the McDonald criteria (both relapse-remitting and progressive)
* Expanded Disability Status Scale (EDSS) score of 2.5 to 6.5 or Patient Determined Disability Score (PDDS) of 2 to 6, indicating preservation of at least some ambulatory function, that is, the ability to walk 20 meters or more, independently, with or without the use of an assistive device
* Willingness to travel to the local study site for the evaluation sessions,
* Internet platform availability

Exclusion Criteria:

* comorbidities hindering participation in the study.
* Individuals who have had a documented relapse and/or corticoid treatment during the past three months will be excluded,
* Individuals with severe cognitive deficits who cannot follow simple instructions and/or consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
30 second sit to stand test | Baseline to 10 weeks
  Measure of lower extremity muscle power and a proxy measure of mobility

SECONDARY OUTCOMES:
Short Physical Performance Battery | Baseline to 10 weeks
  Meaure of balance, walking function and lower extremity muscle strength
Functional Reach Test | Baseline to 10 weeks
  A measure of stability
Timed 25 feet foot walk test | Baseline to 10 weeks
  A measure of walking speed
MiniBESTest | Baseline to 10 weeks
  A measure of balance
Six minute walk test | Baseline to 10 weeks
  A measure of walking endurance
Modified Fatigue Impact Scale | Baseline
  Patient-reported measure of fatigue
12 item Multiple Sclerosis Walking Scale | Baseline to 10 weeks
  Patient-reported outcome of walking function
Multiple Sclerosis Impact Scale | Baseline to 10 weeks
  Patient-reported measure on the impact of multiple sclerosis
EQ-5D-5L | Baseline to 10 weeks
  Patient-reported measure of quality of life
State-Trait Anxiety Inventory | Baseline to 10 weeks
  Patient-reported measure of anxiety
Quick Inventory of Depression Symptomology | Baseline to 10 weeks
  Patient-reported measure of depressive symptoms
Client Services Receipt Inventory | Baseline to 10 weeks
  Patient-reported measure of used health services
Digital Health Literacy Scale | Baseline
  Patient-reported measure of digital health literacy
Telehealth Usability Questionnaire | 10 weeks
  Patient-reported measure of telehealth usability
Semi-structed interview | 10 weeks
  A semi-structured interview on the satisfaction with the telerehabilitation system

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (2):
  - The Danish MS Hospitals, Haslev, Haslev
  - The Danish MS Hospitals, Ry, Ry
- MS Ireland, Dublin, Ireland
- Tel Aviv University, Tel Aviv, Israel
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided